CLINICAL TRIAL: NCT03656523
Title: Management of Antithrombotic TherApy in Patients With Atrial Fibrillation or DevelOping AtRial Fibrillation During Hospitalization for PCI
Acronym: Matador-PCI
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K20
Record Dates: First submitted 2018-08-09; First posted 2018-09-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Coronary Syndrome; Atrial Fibrillation
Keywords: Acute Coronary Syndrome; Atrial Fibrillation; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Coronary Syndrome: Patients with Aute coronary syndrome trated with Percutaneous Coronary Intervention plus Stent implantation and Atrial Fibrillation
  Interventions: Other: Acute coronary syndrome and PCI and AF

INTERVENTIONS:
Other: Acute coronary syndrome and PCI and AF — Patient with ACS and ACS treated with PCI

SUMMARY:
ACS are a potent risk factor for AF, with new onset AF occurring in up to 1 in every 5 patients hospitalized with an ACS.

Despite its relatively frequent occurrence and the many etiologic factors involved in its pathogenetic condition, the frequency and prognostic significance of AF complicating ACS remain unclear

DETAILED DESCRIPTION:
There are limited data available, particularly from a representative population-based perspective describing recent pharmacological and non-pharmacological management and clinical event rates associated with AF complicating ACS in the era of novel treatment strategies (in both AF and ACS) and high coronary reperfusion rates.

This registry will assess the current in-hospital management and clinical events at 6 months of consecutive patients admitted in Italian cardiology intensive care units (CCUs) for an ACS treated invasively with PCI and stent implantation who present AF at admission or during hospital stay, before or after stent implantation .

ELIGIBILITY:
Inclusion Criteria:

* All consecutive ACS patients treated with PCI with stent implantation who present AF at admission or during hospital stay, before or after stent implantation.

Exclusion Criteria:

* Patients admitted with a diagnosis of ACS at the time of enrolment but not confirmed during hospitalization
* ACS treated medically or with PCI but without stent implantation
* Patients not giving informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ACS trated with PCI with stent implantation developing or having Atrial Fibrillation.
Sampling Method: Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Clinical epidemiology | Enrollement
  Demographics
Management | 6 months
  Pharmacological treatment
Antithrombotic strategy | 6 months
  Intravenous or oral antiplatelet and anticoagulation therapies and their combination
Clinical epidemiology | Enrollement
  Clinical history
Clinical epidemiology | Enrollement
  Type of AF
Clinical epidemiology | Enrollement
  Type of ACS
Management | 6 months
  Time of PCI
Number of procedure performed on enrolled patients | 6 months
  In-hospital management

SECONDARY OUTCOMES:
Pharmacological therapies | 6 months
  Use and persistence of therapies prescribed at discharge
Clinical outcomes | 6 months
  All cause deaths, major bleedings, non fatal stroke, systemic embolism, transiet ischemic attach, MI recurrence

CONTACTS AND LOCATIONS:
Locations (76):
- Italy (76):
  - Ospedale Civile Ss. Filippo E Nicola - U.O. Cardiologia E Utic, Avezzano, AQ
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Bari, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Policlinico - U.O. Cardiologia Universitaria, Bari, BA
  - Azienda Ospedaliera G. Rummo - Cardiologia Interventistica E Utic, Benevento, BD
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio, BG
  - Ospedale Civile - Sc Cardiologia, Belluno, BL
  - Ospedale Maggiore - U.O. Di Cardiologia, Bologna, BO
  - Ospedale Nuovo S. Maria Della Scaletta - Uoc Cardiologia, Imola, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Osp. Andria Canosa - Po Andria - Cardiologia - Utic, Andria, BT
  - Azienda Ospedaliera G. Brotzu - Struttura Complessa Di Cardiologia, Cagliari, CA
  - Presidio Ospedaliero Moscati - U.O.C. Cardiologia, Aversa, CE
  - Az. Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia-Utic, Caserta, CE
  - Pineta Grande Hospital - Unita Terapia Intensiva Coronarica, Castel Volturno, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Ospedale Moriggia Pelascini - Unita' Operativa Di Cardiologia, Gravedona, CO
  - Azienda Ospedaliera Cannizzaro - Uoc Cardiologia Con Utic Ed Emodinamica, Catania, CT
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Presidio Ospedaliero T. Masselli Mascia - S.C. Cardiologia - Utic - Riabil. Card., San Severo, FG
  - Ospedale San Giovanni Di Dio - Cardiologia, Florence, FI
  - E.O. Ospedali Galliera - S. C. Cardiologia, Genova, GE
  - Ospedale San Leopoldo Mandic - Cardiologia - Ucc, Merate, LC
  - Ospedale Vito Fazzi - U.O. Di Cardiologia, Lecce, LE
  - Azienda Osp. Cardinale G. Panico - U.O. Cardiologia - Utic, Tricase, LE
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale Di Circolo Di Desio - U.O.C. Di Cardiologia-Utic, Desio, MB
  - Ospedale Civile - Uo Cardiologia, Legnano, MI
  - Ospedale Civile Fornaroli - U.O. Cardiologia, Magenta, MI
  - Centro Cardiologico Monzino - Terapia Intensiva Cardiologica (Utic), Milan, MI
  - Ospedale San Paolo - Uo Cardiologia E Utic, Milan, MI
  - Ospedale San Luca - Istituto Auxologico - U.O. Cardiologia, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia-Ucc, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Ospedale Civile - Unita' Operativa Di Cardiologia, Rho, MI
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Fondazione G. Giglio - U.O. Cardiologia E Utic, Cefalù, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Nuovo Ospedale San Giovanni Battista - S.C. Cardiologia, Foligno, PG
  - Ospedale Di Pordenone - S.O.C. Cardiologia, Pordenone, PN
  - Ospedale Della Val Di Nievole - U. O. Cardiologia - Utic, Pescia, Point
  - Ospedale San Jacopo - U.O. Cardiologia, Pistoia, Point
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Fondazione Irccs Policlinico San Matteo - Card. Con Ucc-Lab. Ricerca Sperim. Card., Pavia, PV
  - Azienda Ospedaliera San Carlo - Ssd Utic, Potenza, PZ
  - Ao Bianchi Melacrino Morelli- Po Riuniti - Divisione Di Cardiologia, Reggio Calabria, RC
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia, RE
  - Ospedale M.P. Arezzo - U.O.C. Cardiologia-Utic, Ragusa, RG
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia 1, Roma, RM
  - Policlinico Umberto Primo - Cardiologia B - Cardiologia E Angiologia, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santo Spirito - U.O.C. Di Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Ospedale Maria Ss. Addolorata - U.O. Di Cardiologia Utic, Eboli, SA
  - Ospedale San Paolo - U.O. Di Cardiologia, Savona, SV
  - Ospedale Santa Maria Del Carmine - Cardiologia, Rovereto, TN
  - Ospedale Santa Chiara - Ospedale Santa Chiara, Trento, TN
  - Ospedale San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Ospedale Degli Infermi - Sc Cardiologia, Rivoli, TO
  - Ospedale Maria Vittoria - U.O. Cardiologia, Torino, TO
  - Ospedale Giovanni Bosco - Sc Cardiologia, Torino, TO
  - Azienda Ospedaliera Santa Maria - S.C. Di Cardiologia, Terni, TR
  - Ospedale Santa Maria Dei Battuti - U.O. Di Cardiologia, Conegliano, TV
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Ospedale Di Circolo E Fondazione Macchi - Ssd Unita' Di Cure Intensive Coronariche, Varese, VA
  - Ospedale Civile - U.O. Cardiologia, Mirano, VE
  - Ospedale Civile - U.O. Cardiologia, San Donà di Piave, VE
  - Casa Di Cura Dr. Pederzoli - Servizio Di Cardiologia, Peschiera del Garda, VR
  - Ospedale Belcolle - U.O.C. Cardiologia Utic Emodinamica, Viterbo, VT
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic, Napoli
  - Pres. Ospedaliero S. Maria Della Pieta' - U.O. Cardiologia E Utic, Nola

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Luca L, Bolognese L, Rubboli A, Vetrano A, Callerame M, Rivetti L, Gonzini L, Gabrielli D, Di Lenarda A, Gulizia MM; MATADOR-PCI Investigators. Combinations of antithrombotic therapies prescribed after percutaneous coronary intervention in patients with acute coronary syndromes and atrial fibrillation: data from the nationwide MATADOR-PCI registry. Eur Heart J Cardiovasc Pharmacother. 2021 May 23;7(3):e45-e47. doi: 10.1093/ehjcvp/pvaa088. No abstract available. PMID 32651996
- [Result] De Luca L, Rubboli A, Bolognese L, Gonzini L, Urbinati S, Murrone A, Scotto di Uccio F, Ferrari F, Luca F, Caldarola P, Lucci D, Gabrielli D, Di Lenarda A, Gulizia MM; MATADOR-PCI Investigators. Antithrombotic management of patients with acute coronary syndrome and atrial fibrillation undergoing coronary stenting: a prospective, observational, nationwide study. BMJ Open. 2020 Dec 22;10(12):e041044. doi: 10.1136/bmjopen-2020-041044. PMID 33371033